CLINICAL TRIAL: NCT06956235
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Tulisokibart in Participants With Moderate to Severe Hidradenitis Suppurativa
Brief Title: Study to Evaluate Tulisokibart for Hidradenitis Suppurativa (MK-7240-012)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7240-012; U1111-1316-5263 (Registry Identifier: UTN); 2024-520039-33-00 (Registry Identifier: EU CT); jRCT2011250007 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); MK-7240-012 (Other: MSD)
Record Dates: First submitted 2025-04-30; First posted 2025-05-04 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1: High Dose (Experimental): Participants receive a high dose tulisokibart regimen.
  Interventions: Drug: Tulisokibart
- Arm 2: Medium Dose (Experimental): Participants receive a medium dose tulisokibart regimen.
  Interventions: Drug: Tulisokibart
- Arm 3: Low Dose (Experimental): Participants receive a low dose tulisokibart regimen.
  Interventions: Drug: Tulisokibart
- Arm 4: Placebo (Placebo Comparator): Participants receive a placebo regimen, and are then allocated to a medium or high tulisokibart dose regimen after Week 16.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tulisokibart — Solution in autoinjector for subcutaneous (SC) injection
  Other Names: PRA023; MK-7240
  Arms: Arm 1: High Dose; Arm 2: Medium Dose; Arm 3: Low Dose
Drug: Placebo — Solution in autoinjector for SC injection
  Arms: Arm 4: Placebo

SUMMARY:
This is a phase 2b randomized, double-blind, placebo-controlled study of the safety and efficacy of tulisokibart in participants with moderate to severe hidradenitis suppurativa. The primary hypothesis is that at least 1 dose of tulisokibart is superior to placebo with respect to the proportion of participants achieving a 50% reduction in Hidradenitis Suppurativa Clinical Response (HiSCR50) at Week 16 (ie, at end of double-blind treatment).

DETAILED DESCRIPTION:
This study consists of a 16-week Double-blind Period and a 100-week Long-term Extension (LTE) composed of a 40-week Main Extension and a 60-week Optional Extension.

ELIGIBILITY:
Inclusion Criteria:

* Has signs and symptoms of hidradenitis suppurativa (HS) for ≥6 months prior to Screening and a clinical diagnosis of HS at Screening
* Has moderate or severe HS defined as a total combined number of ≥ 5 abscesses and/or inflammatory nodules, with HS lesions present in ≥ 2 distinct anatomical areas and ≥ 1 anatomic area of HS involvement characterized as Hurley Stage II or III
* Has a history of inadequate response to a course of systemic antibiotics for treatment of HS or intolerance to or has a contraindication to systemic antibiotics for treatment of HS
* Has ≤20 draining tunnel count at Screening and Randomization

Exclusion Criteria:

* Has other active skin conditions that may, in the judgment of the investigator, interfere with the assessment of HS
* Has any immune-mediated inflammatory condition that is not well controlled and which may potentially require biologic therapy
* Has a transplanted organ and requires continued systemic immunosuppression
* Has a history of cancer (except fully treated nonmelanoma skin cancers or cervical carcinoma in situ after complete surgical removal) and is disease free for <5 years
* Has had a diagnostic evaluation suggestive of malignancy (eg, chest or breast imaging) and the possibility of malignancy cannot be reasonably excluded following additional clinical assessments
* Has a known infection with hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV)
* Has any active infection
* Has active tuberculosis
* Has had major surgery within the past 3 months or has a major surgery planned during the study
* Has a history of clinically significant drug or alcohol abuse within the past 6 months
* Has prior exposure to tulisokibart
* Has undergone laser therapy or surgical procedures for their lesions within the past 6 weeks or is planning to have laser therapy or surgical procedures for lesions during participation in the study
* Has known allergies, hypersensitivity, or intolerance to tulisokibart or its excipients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2026-11-16 (Estimated); Study Completion 2029-01-22 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Hidradenitis Suppurativa Clinical Response (HiSCR) 50 at Week 16 | Week 16
  The percentage of participants with ≥50% reduction in total abscesses and inflammatory nodules (AN) count with no increase in abscess count, and no increase in draining tunnels (ie, HiSCR50) will be reported.

SECONDARY OUTCOMES:
Percentage of Participants Achieving HiSCR75 at Week 16 | Week 16
  The percentage of participants with ≥75% reduction in total abscesses and inflammatory nodules (AN) count with no increase in abscess count, and no increase in draining tunnels (ie, HiSCR75) will be reported.
Mean Change from Baseline in Dermatology Life Quality Index (DLQI) at Week 16 | Week 16
  The DLQI is a validated dermatology-specific instrument that measures the HRQoL in adult patients with skin diseases. The DLQI consists of 10 questions and provides a total HRQoL score, as well as scores for 6 aspects of QoL: symptoms and feelings; daily activities; leisure; work/school; personal relationships; and treatment. The recall period is over the last week. Question responses are assessed using a 4-point Likert rating scale ranging from "not at all" (scored 0) to "very much" (scored 3). The final score ranges from 0 (no impact on QOL) to 30 (maximum impairment). The mean change from baseline in DLQI at Week 16 will be reported.
Percentage of Participants Who Experience One or More Adverse Events (AEs) | Up to ~130 weeks
  An AE is defined as any untoward medical occurrence in a participant administered a study treatment which did not necessarily have to have a causal relationship with this treatment. An AE could be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of study treatment, is also an AE. The percentage of participants with any AE will be reported.
Percentage of Participants Who Discontinue Study Intervention Due to an AE | Up to ~116 weeks
  An AE is defined as any untoward medical occurrence in a participant administered a study treatment which did not necessarily have to have a causal relationship with this treatment. An AE could be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of study treatment, is also an AE. The percentage of participants discontinuing from study intervention due to AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (68):
- United States (19):
  - Cahaba Dermatology & Skin Health Center ( Site 0012), Birmingham, Alabama
  - Medical Dermatology Specialists ( Site 0027), Phoenix, Arizona
  - Northwest Arkansas Clinical Trials Center, PLLC ( Site 0049), Rogers, Arkansas
  - Northridge Clinical Trials ( Site 0004), Northridge, California
  - Integrative Skin Science and Research ( Site 0015), Sacramento, California
  - Olympian Clinical Research ( Site 0010), Tampa, Florida
  - Skin Care Physicians of Georgia ( Site 0033), Macon, Georgia
  - Dawes Fretzin Clinical Research Group, LLC ( Site 0025), Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center ( Site 0044), Boston, Massachusetts
  - Revival Research Institute, LLC ( Site 0005), Troy, Michigan
  - Mount Sinai Doctors - East 85th Street ( Site 0050), New York, New York
  - DJL Clinical Research, PLLC ( Site 0021), Charlotte, North Carolina
  - University Hospitals Cleveland Medical Center ( Site 0046), Cleveland, Ohio
  - Wright State Physicians Health Center ( Site 0041), Fairborn, Ohio
  - Palmetto Clinical Trial Services, LLC ( Site 0023), Anderson, South Carolina
  - Arlington Center for Dermatology ( Site 0045), Arlington, Texas
  - Texas Dermatology Research Center ( Site 0019), Dallas, Texas
  - Reveal Research Institute ( Site 0018), Frisco, Texas
  - Progressive Clinical Research ( Site 0020), San Antonio, Texas
- Argentina (4):
  - CIPREC ( Site 0202), CABA
  - Hospital Italiano de Buenos Aires ( Site 0205), CABA
  - Psoriahue ( Site 0203), CABA
  - Derma Internacional SA ( Site 0206), CABA
- Australia (3):
  - Liverpool Hospital ( Site 1403), Liverpool, New South Wales
  - The Alfred Hospital ( Site 1401), Melbourne, Victoria
  - Fremantle Dermatology ( Site 1402), Fremantle, Western Australia
- Canada (5):
  - Wiseman Dermatology Research Inc. ( Site 0107), Winnipeg, Manitoba
  - Brunswick Dermatology Center ( Site 0101), Frederiction, New Brunswick
  - Lynderm Research Inc. ( Site 0104), Markham, Ontario
  - SKiN Centre for Dermatology ( Site 0103), Peterborough, Ontario
  - York Dermatology Clinic & Research Centre ( Site 0106), Richmond Hill, Ontario
- Chile (3):
  - Centro Skin Med Limitada ( Site 0305), Santiago, Region M. de Santiago
  - Clinica Dermacross ( Site 0301), Santiago, Region M. de Santiago
  - Centro Internacional de Estudios Clinicos (CIEC) ( Site 0302), Santiago, Region M. de Santiago
- China (7):
  - Dermatology Hospital of Southern Medical University ( Site 1504), Guangzhou, Guangdong
  - The Second Xiangya Hospital of Central South University ( Site 1505), Changsha, Hunan
  - The First Hospital of Jilin University ( Site 1502), Changchun, Jilin
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine ( Site 1515), Shanghai, Shanghai Municipality
  - Huashan Hospital of Fudan University ( Site 1506), Shanghai, Shanghai Municipality
  - PEOPLE'S HOSPITAL OF XINJIANG UYGUR AUTONOMOUS REGION ( Site 1509), Ürümqi, Xinjiang
  - The first Affiliated Hospital, Zhejiang University School of Medicine ( Site 1501), Hangzhou, Zhejiang
- Colombia (2):
  - Servicios de Salud IPS Suramericana S.A.S. - IPS Sura San Diego ( Site 0404), Medellín, Antioquia
  - Fundación Valle del Lili ( Site 0403), Cali, Valle del Cauca Department
- France (4):
  - Hôpital Edouard Herriot ( Site 0601), Lyon, Auvergne-Rhône-Alpes
  - CHU de Bordeaux Hop St ANDRE ( Site 0603), Bordeaux, Gironde
  - HIA Sainte Anne ( Site 0606), Toulon, Var
  - Hopitaux Universitaires Paris Centre-Hopital Cochin ( Site 0602), Paris
- Germany (2):
  - Frankfurt Universitaetsklinikum EC ( Site 0706), Frankfurt am Main, Hesse
  - Charite - Universtitatsmedizin Berlin CCM ( Site 0708), Berlin
- Italy (3):
  - AOU Ospedali Riuniti di Ancona ( Site 1805), Ancona, The Marches
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico ( Site 1806), Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore ( Site 1801), Roma
- Japan (6):
  - Nagoya City University Hospital ( Site 1603), Nagoya, Aichi-ken
  - Medical Corporation Kojinkai Sapporo Skin Clinic ( Site 1606), Sapporo, Hokkaido
  - University of the Ryukyus Hospital ( Site 1601), Ginowan, Okinawa
  - Nihon University Itabashi Hospital ( Site 1602), tabashi City, Tokyo
  - Fukuoka University Hospital ( Site 1604), Fukuoka
  - University Hospital,Kyoto Prefectural University of Medicine ( Site 1605), Kyoto
- Netherlands (2):
  - Amphia Ziekenhuis, locatie Breda Molengracht ( Site 0902), Breda, North Brabant
  - Erasmus Medisch Centrum ( Site 0901), Rotterdam, South Holland
- Singapore (2):
  - National Universtity Hospital IMU ( Site 0802), Singapore, Central Singapore
  - National Skin Centre ( Site 0801), Singapore, Central Singapore
- Spain (4):
  - Hospital de Manises ( Site 1103), Manises, Valencia
  - Hospital Universitari Vall d'Hebron ( Site 1102), Barcelona
  - Hospital Universitari de Bellvitge ( Site 1101), Barcelona
  - Hospital Universitario Virgen Nieves ( Site 1104), Granada
- United Kingdom (2):
  - Russells Hall Hospital ( Site 1303), Dudley, England
  - Royal London Hospital ( Site 1301), London, England

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com